CLINICAL TRIAL: NCT02426151
Title: A Randomized, Open Label, Single-dose 2x2 Crossover Study to Compare Pharmacokinetic, Pharmacodynamic Profiles, and Tolerability of EPO (BEPO-A (4000 IU)) and EPO (REPO-A (4000 IU)) in Healthy Male Subjects
Brief Title: Bioequivalence of a Single Subcutaneous Dose of BEPO and REPO in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-EPCL009
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2015-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BEPO-A (Experimental): Single subcutaneous injection of BEPO-A 4000 IU (Bioreactor manufacturing process)
  Interventions: Drug: BEPO-A
- REPO-A (Active Comparator): Single subcutaneous injection of REPO-A 4000 IU (Roller bottle manufacturing process)
  Interventions: Drug: REPO-A

INTERVENTIONS:
Drug: BEPO-A — BEPO-A (Bioreactor manufacturing process)
  Arms: BEPO-A
Drug: REPO-A — REPO-A (Roller bottle manufacturing process)
  Arms: REPO-A

SUMMARY:
To Compare Pharmacokinetic and Pharmacodynamic Profiles of BEPO-A and REPO-A in Healthy Male Subjects

DETAILED DESCRIPTION:
To Compare Pharmacokinetic and Pharmacodynamic Profiles of EPO (BEPO-A (4000 IU)) and EPO (REPO-A (4000 IU)) in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Agree to all the purposes of the study by signing and dating the Informed Consent;
* Male, aged between 19 and 40 years, clinically healthy;
* BMI between 19 and 28;
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP < 85 mmHg

Exclusion Criteria:

* Hemoglobin <13 g / dL
* Ferritin <20 ng/mL or TIBC > 360 ug/ dL
* Vitamin B12 < 200 pg/mL or floate < 4 ng/mL
* %reticulpcyte > 3%
* platelet < 100,000/ul or > 400,000/ul
* GFR < 60mL/min/1.73m2
* Going to or during treatment of the tumor
* Clinical history of allergy of biological products derived from mammalian albumin or any component of the formulation
* Clinical history of autoimmune or hereditary anemia
* A Positive reaction in the nicotine tests
* Principal Investigator of the study criteria.

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cmax and AUClast | 1D before dosing, 1h, 2, 4h, 7h, 10h,12h, 14h, 2D 0h, 2D 8h, 3D 0h, 4D 0h, 5D 0h, 6D 0h,

SECONDARY OUTCOMES:
AUCinf, Tmax, t1/2β, CL/F, MRTinf (mean residence time) of Erythropoietin | 1D before dosing, 1h, 2, 4h, 7h, 10h,12h, 14h, 2D 0h, 2D 8h, 3D 0h, 4D 0h, 5D 0h, 6D 0h,

IPD SHARING:
Plan to Share IPD: No